CLINICAL TRIAL: NCT06800911
Title: Metacognitive Beliefs, Emotional Regulation in Obese Patients
Brief Title: Metacognitive Beliefs in Obese Patients
Acronym: METAOBES
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C415
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: Metabeliefs; Metacognition; Rumination; Dysfunctional lifestyle; Rehabilitation
MeSH Terms: conditions — Obesity; Rumination Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obesity: Patients aged between 18 and 65, of both sexes, of Italian nationality, suffering from obesity (Body Mass Index, BMI: kg/m2 ≥ 35, according to the criteria of the World Health Organization WHO).
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Metacognition Questionnaire Penn State Worry Questionnaire Ruminative Response Scale Anger Rumination scale Difficulties in Emotion Regulation Scale Emotional Eating subscale of the Dutch Eating Behavior Questionnaire

SUMMARY:
The study aims to investigate the presence of metacognitive beliefs, emotional regulation, and emotional eating in obese patients and their possible relationships.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 65 years
* Italian nationality
* Body Mass Index ≥ 35 kg/m2

Exclusion Criteria:

* Psychiatric pathologies
* Severe cognitive deficits that could compromise the completion of the questionnaires
* Absence of signed informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 90 patients aged between 18 and 65, of both sexes, of Italian nationality, suffering from obesity (Body Mass Index, BMI: kg/m2 ≥ 35, according to the criteria of the World Health Organization WHO).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Metacognitive beliefs | Baseline
  Metacognition Questionnaire (MCQ-30) is a self-report test composed of 30 items on a 4-point Likert scale from 1 (I do not agree) to 4 (I completely agree agreement).
Rumination | Baseline
  Ruminative Response Scale (RRS) is a self-report test composed of 20 items on a 4-point Likert scale from 1 (almost never) to 4 (almost always).
Anger Rumination | Baseline
  Anger Rumination scale (ARS) is a self-report test composed of 14 items, on a Likert scale from 1 (almost never) to 4 (almost always).
Emotional dysregulation | Baseline
  Difficulties in Emotion Regulation Scale (DERS) isa self-report test composed of 36 items on a Likert scale from 1 (almost never) to 5 (almost always).
Emotional eating | Baseline
  Emotional Eating subscale of the Dutch Eating Behavior Questionnaire (DEBQ), composed of 13 items on a Likert scale from 0 (never) to 4 (almost always)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy